CLINICAL TRIAL: NCT01112735
Title: A Randomized, Controlled, Multicenter Phase 2 Study to Evaluate the Efficacy and Safety of ARTISS (FS VH S/D 4 S-apr) for Flap Adherence in Subjects Undergoing Abdominoplasty
Brief Title: Efficacy and Safety of ARTISS for Flap Adherence in Abdominoplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 550902
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Seroma; Hematoma
Keywords: Abdominoplasty; Flap adherence in subjects undergoing abdominoplasty to eliminate dead space and reduce seroma/hematoma formation
MeSH Terms: conditions — Seroma; Hematoma | interventions — Low Density Lipoprotein Receptor-Related Protein-1; Standard of Care

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- ARTISS (Experimental): ARTISS will be used as an adjuvant to standard of care.
  Interventions: Biological: FS VH S/D 4 s-apr (= two-component fibrin sealant, double virus inactivated, made from pooled human plasma)
- Standard of care (Other): Standard of care
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Biological: FS VH S/D 4 s-apr (= two-component fibrin sealant, double virus inactivated, made from pooled human plasma) — Dosage form: spray (aerosolized sealant), Dosage frequency: once (1 layer). ARTISS will be applied onto the fascia or the wound bed.
  Other Names: ARTISS
  Arms: ARTISS
Procedure: Standard of care — Standard of care
  Arms: Standard of care

SUMMARY:
The purpose of the study is to compare the safety and efficacy of ARTISS versus standard of care in adhering tissue places and reducing seroma/hematoma formation in subjects undergoing abdominoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 75 years of age at the time of screening
* Subject is planned for primary standard abdominoplasty (status post Cesarean section or liposuction performed more than 6 months prior to enrollment in the study are allowed)
* If the subject is of childbearing potential; presents with a negative pregnancy test, and agrees to employ adequate birth control measures for the duration of the study
* Subject resides within 100 miles of the investigational site and is willing and able to comply with the scheduling requirements of the protocol (notably home visits by study personnel)
* Subject is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Subject is obese (body mass index [BMI] > 30 before surgery)
* Subject has experienced massive weight loss (subject has a history of obesity during adult life; subject lost more than 20 BMI unit score, subject has undergone a bariatric surgery)
* Subject has a history of active smoking within the previous 12 months
* Subject is elected for a non-standard abdominoplasty (extended, limited or mini-abdominoplasty, endoscopic, fleur-de-lis or circumferential abdominoplasty) or panniculectomy
* Subject has scars on the abdominal wall above the umbilicus. Vertical midline, laparoscopic punctures, or liposuction punctures are permitted
* Subject is planned for other "body lifting" procedures (eg to the arms, legs, back etc.)
* Subject is planned for combined abdominoplasty with other cosmetic procedures including liposuction (restricted liposuction of the waist line and the lower back is allowed, as long as the integrity of the surgical spaces is maintained)
* Subject has an active or chronic skin disorder, history or evidence of keloid formation, or hypertrophic scarring
* Subject has a history of gastrointestinal disorders (eg Irritable Bowel Syndrome) requiring prescription medications
* Subject has a known abdominal hernia that requires mesh fixation
* Subject has a documented hiatal hernia or acid reflux disease
* Subjects with congenital or acquired immunodeficiency disorders
* Subject has uncontrolled diabetes mellitus (HbA1c > 7.0)
* Subject has a history of cardio-vascular disease including uncontrolled hypertension (> 140/90 mm Hg)
* Subject has a clinically diagnosed psychiatric disorder (including obsessive compulsive disorders)
* Subject has a known (documented) bleeding or coagulation disorder including history of thromboembolic events
* Subject is being treated with anti-coagulants or with Aspirin (that was not discontinued 7 days prior to surgery)
* Subject is receiving active treatment for a malignancy
* Subject has a connective tissue disorder
* Subject has received chronic treatment with immunosuppressive drugs, systemic corticosteroids, or other chronic treatments within 30 days prior to the surgery
* Subject has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study
* Subject has a known sensitivity to fibrin sealants
* Subject is a friend, employee, or relative of the investigator or other study personnel

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Z Abrams, MD, MBA, Study Director — Baxter Healthcare Corporation
Locations (6):
- United States (6):
  - Mei Li Surgery Center, Beverly Hills, California
  - Center for Plastic Surgery and Skin Care, Fort Lauderdale, Florida
  - Miami Plastic Surgery, Miami, Florida
  - Places Plastic Surgery, Atlanta, Georgia
  - The Practice of Gary Wiesman, M.D. and Irvin Wiesman, M.D. and Associates, Chicago, Illinois
  - UT Southwestern Medical Center, Department of Plastic Surgery, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- ARTISS: ARTISS will be used as an adjuvant to standard of care.
  ARTISS, also known as "FS VH S/D 4 s-apr" is a Fibrin Sealant Vapor Heated Solvent/Detergent Treated, and is a double virus inactivated 2-component fibrin sealant made from pooled human plasma.
  The dosage form is spray (aerosolized sealant) in a 10mL kit, and frequency was once (1 layer) applied at a dosing volume of between 0.02mL/cm2 and 0.04 mL/cm2 onto the fascia or the wound bed. The fibrin sealant matrix is biodegradable and disappears over a 2-3 week period.
Period: Overall Study
Arm/Group | ARTISS | Standard of Care
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARTISS | Standard of Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.90 (7.89) | 45.60 (10.32) | 43.25 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 14 | 13 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 20 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Drainage Volume Collected Until Drain Removal
Description: Drainage fluids were to be collected through the Blake drain and into the collection bulb. The drainage volume was measured and recorded daily until the removal of the drain. During scheduled visits, measurement was to be performed at the study site, and on non-visit day recording of the drainage volume was to be done by a visiting home care nurse (or other study personnel). The drain was ready to be removed when the drainage volume in a given 24 hour period was <=30 cc.
Time Frame: Day 0 (Surgery Day) to Day 90
Population: Full Analysis Set (FAS) consists of all subjects who were randomized (ie, the investigator opened the randomization envelope) and treated and who had an available assessment for the primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | ARTISS | Standard of Care
Number analyzed (Participants) | 20 | 20
mL | 407.45 (470.36) | 595.90 (519.46)

2. Secondary Outcome: Occurrence of Seroma
Description: The investigator inspected each subject post surgery (Day 0) an each scheduled visit (Day 3, 7, 14, 28, 60, 90) to determine whether there were any areas on the abdominal wall that meet the definition of seroma. A seroma is a pocket of clear serous fluid that sometimes develops in the body after surgery. This fluid is composed of blood plasma that has seeped out of ruptured small blood vessels and inflammatory fluid produced by the injured and dying cells.
Time Frame: Day 0 (Surgery Day) to Day 90
Population: FAS
Measure: Number; unit: Events
Arm/Group | ARTISS | Standard of Care
Number analyzed (Participants) | 20 | 20
Events | 8 | 5

3. Secondary Outcome: Occurrence of Hematoma
Description: The investigator inspected each subject post surgery (Day 0) an each scheduled visit (Day 3, 7, 14, 28, 60, 90) to determine whether there were any areas on the abdominal wall that meet the definition of hematoma. A hematoma is a collection of blood outside of a blood vessel.
Time Frame: Day 0 (Surgery Day) to Day 90
Population: FAS
Measure: Number; unit: Events
Arm/Group | ARTISS | Standard of Care
Number analyzed (Participants) | 20 | 20
Events | 0 | 0

4. Secondary Outcome: Time to Drain Removal
Description: The drain was ready to be removed when the drainage volume in a given 24 hour period was <=30cc.
Time Frame: Day 0 (Surgery Day) up to Day 90
Population: FAS
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ARTISS | Standard of Care
Number analyzed (Participants) | 20 | 20
Days | 6.8 (7.11) | 9.55 (5.82)

5. Secondary Outcome: Number of Fluid Aspiration for Seromas
Description: Number of interventions recorded.
Time Frame: Day 0 (Surgery Day) to Day 90
Population: FAS
Measure: Mean (Standard Deviation); unit: Interventions
Arm/Group | ARTISS | Standard of Care
Number analyzed (Participants) | 8 | 5
Interventions | 5 (4.34) | 3.2 (1.64)
Statistical Analysis 1: Comparison: ARTISS vs Standard of Care; Test type: Superiority; p = 0.5621, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Total Volume of Fluid Aspirations for Seromas
Description: Volume of fluid recovered was recorded.
Time Frame: Day 0 (Surgery Day) to Day 90
Population: FAS
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | ARTISS | Standard of Care
Number analyzed (Participants) | 8 | 5
mL | 226.13 (157.78) | 152.2 (150.34)
Statistical Analysis 1: Comparison: ARTISS vs Standard of Care; Test type: Superiority; p = 0.3595, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change From Baseline in Postoperative Skin Sensitivity 2 Inches Above Umbilicus
Description: Test administered on abdomen midline using a set of different size Semmes-Weinstein monofilaments. These instruments are used to measure the cutaneous sensory perception threshold of patients. Each monofilament represents a unique amount of force. The force applied by each monofilament increases with each ascending size. Testing begins with small to large monofilaments. A higher score indicates a greater loss of sensation. Evaluator Size=ES, Hand & Dorsal Foot Thresholds=HDFT, Normal=N, Diminished Light Touch=DLT,Diminished Protective Sensation=DPS, Loss of Protective Sensation=LOPS, Deep Pressure Sensation Only=DPSO:
  ES=1.65 (minimum),HDFT=N;ES=2.36,HDFT=N;ES=2.44,HDFT=N;ES=2.83,HDFT=N;ES=3.22,HDFT=DLT;ES=3.61,HDFT=DLT;ES=3.84,HDFT=DPS;ES=4.08,HDFT=DPS;ES-4.17,HDFT=DPS;ES=4.31,HDFT=DPS;ES=4.56,HDFT=LOPS;ES=4.74,HDFT=LOPS;ES=4.93,HDFT=LOPS;ES=5.07,HDFT=LOPS;ES=5.18,HDFT=LOPS;ES=5.46,HDFT=LOPS;ES=5.88,HDFT=LOPS;ES=6.10,HDFT=LOPS;ES=6.45,HDFT=LOPS;ES=6.65 (maximum),HDFT=DPSO.
Time Frame: Days 0 (Baseline), 3, 7, 14, 28, 60, 90
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ARTISS | Standard of Care
Number analyzed (Participants) | 20 | 20
Units on a Scale
  Day 3 | 0.92 (1.79) | 0.89 (1.69)
  Day 7 | 0.55 (1.37) | 0.73 (1.34)
  Day 14 | 0.78 (1.42) | 0.54 (1.08)
  Day 28 | 0.63 (1.41) | 0.53 (1.28)
  Day 60 | 0.5 (1.26) | 0.3 (1.46)
  Day 90 | 0.38 (0.95) | 0.19 (1.17)
Statistical Analysis 1: Comparison: ARTISS vs Standard of Care; Day 3; Test type: Superiority; p = 0.9417, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ARTISS vs Standard of Care; Day 7; Test type: Superiority; p = 0.5488, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ARTISS vs Standard of Care; Day 14; Test type: Superiority; p = 0.7107, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: ARTISS vs Standard of Care; Day 28; Test type: Superiority; p = 0.8809, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: ARTISS vs Standard of Care; Day 60; Test type: Superiority; p = 0.4598, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: ARTISS vs Standard of Care; Day 90; Test type: Superiority; p = 0.3837, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change From Baseline in Postoperative Skin Sensitivity 1 Inch Below Umbilicus
Description: Test administered on abdomen midline using a set of different size Semmes-Weinstein monofilaments. These instruments are used to measure the cutaneous sensory perception threshold of patients. Each monofilament represents a unique amount of force. The force applied by each monofilament increases with each ascending size. Testing begins with small to large monofilaments, pressing at a 90 degree angle for approximately 1.5 seconds against the skin until it bows then it is removed. The patient is instructed to respond when a stimuli is felt, and a score is applied based on the monofilament in use. A higher score indiactes a greater loss of sensation.
Time Frame: Days 0 (Baseline), 3, 7, 14, 28, 60, 90
Population: FAS
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | ARTISS | Standard of Care
Number analyzed (Participants) | 20 | 20
Score on a Scale
  Day 3 | 1.81 (1.83) | 1.78 (1.67)
  Day 7 | 1.47 (1.32) | 1.02 (1.52)
  Day 14 | 1.28 (1.47) | 0.49 (1.25)
  Day 28 | 1.21 (1.43) | 0.81 (1.45)
  Day 60 | 0.97 (1.67) | 0.50 (1.55)
  Day 90 | 1.00 (1.68) | 0.84 (1.42)
Statistical Analysis 1: Comparison: ARTISS vs Standard of Care; Day 3; Test type: Superiority; p = 0.9699, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ARTISS vs Standard of Care; Day 7; Test type: Superiority; p = 0.4709, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ARTISS vs Standard of Care; Day 14; Test type: Superiority; p = 0.1406, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: ARTISS vs Standard of Care; Day 28; Test type: Superiority; p = 0.4291, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: ARTISS vs Standard of Care; Day 60; Test type: Superiority; p = 0.2704, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: ARTISS vs Standard of Care; Day 90; Test type: Superiority; p = 0.7564, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Summary of Pain Assessment by Visit
Description: Subjects were to be presented with a non-verbal visual analogue scale (VAS) to measure the level of pain (rating 0 [no pain] to 10 [worst possible pain]) the patient experienced at the site of surgery at the time of the visit.
Time Frame: Day 3, 7, 14, 28, 60, 90
Population: FAS
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | ARTISS | Standard of Care
Number analyzed (Participants) | 20 | 20
Score on a Scale
  Day 3 | 3.68 (2.40) | 4 (2.03)
  Day 7 | 2.7 (2.11) | 2.8 (1.79)
  Day 14 | 1.7 (1.53) | 1.7 (1.34)
  Day 28 | 1.05 (1.73) | 0.37 (0.50)
  Day 60 | 0.37 (0.76) | 0.3 (0.57)
  Day 90 | 0.3 (0.92) | 0.15 (0.37)

10. Secondary Outcome: Summary of Numbness Assessment by Visit
Description: Subjects were to be presented with a non-verbal VAS to measure the level of numbness (rating 0 [no numbness] to 10 [complete numbness]) that the patient experienced at the time of the visit.
Time Frame: Day 3, 7, 14, 28, 60, 90
Population: FAS
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | ARTISS | Standard of Care
Number analyzed (Participants) | 20 | 20
Score on a Scale
  Day 3 | 5.16 (3.24) | 6.30 (2.39)
  Day 7 | 5.50 (2.54) | 4.95 (2.21)
  Day 14 | 4.45 (2.52) | 4.35 (2.32)
  Day 28 | 3.25 (1.92) | 3.42 (2.61)
  Day 60 | 3.37 (1.74) | 3.16 (2.29)
  Day 90 | 2.85 (1.69) | 2.11 (1.91)

ADVERSE EVENTS:
Time Frame: 90 days
Description: An AE was defined as any untoward medical occurrence in a subject administered IP that does not necessarily have a causal relationship with the treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an IP, whether or not related to the IP. An AE included any event, regardless of the presumed causality between the event and the IP.
Arm/Group | ARTISS | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 10/20 | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARTISS (N=20) | Standard of Care (N=20)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARTISS (N=20) | Standard of Care (N=20)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incision Site Infection (Infections and infestations) | 1 (1) | 1 (1)
Abdominal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 8 (9) | 5 (6)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Staphylococcus Test Positive (Investigations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Incision Site Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes